CLINICAL TRIAL: NCT06988956
Title: A Prospective, Randomized Controlled, Open Label, Multicenter, Phase II Clinical Study Evaluating the Efficacy and Safety of Nimotuzumab Combined With Concurrent Chemoradiotherapy in Elderly Patients With Locally Advanced Unresectable Esophageal Squamous Cell Carcinoma
Brief Title: Nimotuzumab Plus Definite Chemoradiotherapy(dCRT) in Elderly Patients With Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ge Xiaolin, Clinical Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IST-Nim-ESCC-23
Record Dates: First submitted 2024-04-01; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Nimotuzumab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — nimotuzumab; Tegafur; S 1 (combination); Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nimotuzumab plus concurrent chemoradiotherapy group (Experimental): S-1: TBSA<1.4 m²，40mg；TBSA=1.4-1.6 m²，50mg；TBSA>1.6 m²，60mg,po,BID, During the synchronous period of radiotherapy，QW，D1-D5, After radiotherapy，Q3W，D1-14，lasting for 1 year Nimotuzumab 400mg, iv, D1, Week 1; Nimotuzumab 200mg, iv, D8, QW, weeks 2-5. The prescribed dose required 95％PTV 50.4Gy/1.8Gy/28f SIB-PGTV 59.92Gy/2.14Gy/28 次
  Interventions: Drug: Nimotuzumab; Drug: Tegafur; Radiation: radiotherapy
- concurrent chemoradiotherapy group alone (Active Comparator): S-1: TBSA<1.4 m²，40mg；TBSA=1.4-1.6 m²，50mg；TBSA>1.6 m²，60mg,po,BID, During the synchronous period of radiotherapy，QW，D1-D5, After radiotherapy，Q3W，D1-14，lasting for 1 year The prescribed dose required 95％PTV 50.4Gy/1.8Gy/28f SIB-PGTV 59.92Gy/2.14Gy/28 次
  Interventions: Drug: Tegafur; Radiation: radiotherapy

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab 400mg
  Other Names: Nim
  Arms: Nimotuzumab plus concurrent chemoradiotherapy group
Drug: Tegafur — S-1 60mg/m2
  Other Names: S-1
Radiation: radiotherapy — PTV 50Gy/2Gy

SUMMARY:
investigators plan to conduct a multicenter, prospective, randomized controlled, open, phase clinical study to compare the efficacy and safety of nimotuzumab with concurrent chemoradiation alone in elderly participants with advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
investigators plan to conduct a multicenter, prospective, randomized controlled, open, phase clinical study to compare the efficacy and safety of nimotuzumab with concurrent chemoradiation alone in elderly participants with advanced esophageal squamous cell carcinoma. The enrolled participants will be randomly ized into the trial and control group according to 1:1. The test group received nimotuzumab and radiotherapy; the control group received Tigio and radiotherapy. This study includes the screening period, treatment period, efficacy follow-up period, and survival follow-up period

ELIGIBILITY:
Inclusion Criteria:

1. The subject volunteered to join the study, signed the informed consent form, had good compliance, and cooperated with the follow-up;
2. Age 70 or above, male or female;
3. The ECOG score is 0-1 point;
4. Oesophageal squamous cell carcinoma diagnosed by histology or cytology;
5. According to the efficacy evaluation criteria of solid tumors (RECIST 1.1), at least one measurable lesion, and the measurable lesion should not receive local treatment such as radiotherapy (the lesion located in the previous radiotherapy area can also be selected if the progression is confirmed and meets the RECIST1.1 criteria);
6. Stage II-IVB (IVB stage only includes supraclavicular/abdominal lymph node metastasis, does not include any other distant metastasis), can tolerate synchronous radiotherapy, chemotherapy, and targeted therapy
7. Expected survival time of 6 months;
8. Main organ function is normal, that is, meet the following criteria:

1) Blood routine examination:

1. HBG≥90g/L；
2. ANC≥1.5×109/L；
3. PLT ≥80×109/L； 2) Biochemical examination:

a.ALB≥30g/L； B. ALT and AST≤2.5ULN; ALT and AST 5 ULN; c.TBIL≤1.5ULN； D. Plasma Cr≤1.5ULN or creatinine clearance (CCr) of 60 ml/min; 9. Echocardiographic assessment: left ventricular ejection fraction (LVEF) low normal value (50%); 10. Women of childbearing age should agree to use contraception (e. g. intrauterine devices, contraceptives or condoms) during the study and within 6 months after the study; serum or urine pregnancy tests were negative within 7 days before study enrollment and must be non-lactating patients; men who agree to use contraception during the study and within 6 months after the end of the study period.

Exclusion Criteria:

1. Received EGFR mAb and EGFR-TKI within half a year;
2. Participated in other interventional clinical trials within 30 days before screening;
3. Have serious concurrent diseases, such as heart failure, high risk of uncontrolled arrhythmia, severe myocardial infarction, intractable hypertension, renal failure (CKD-4 and above), thyroid insufficiency, mental illness, diabetes, severe chronic diarrhea (more than 7 times a day) and the researchers think not suitable to participate in the clinical research;
4. Patients with brain metastases with symptoms or symptom control time for less than 3 months;
5. History of other malignant tumors (except for cured cervical carcinoma in situ or basal cell carcinoma of the skin and other malignant tumors that have been cured for more than 5 years);
6. presence of active infection or active infectious diseases;
7. The presence of multilevel esophageal malignancy or signs of esophageal fistula and perforation;
8. Patients whose imaging shows that the tumor has invaded important blood vessels or whose tumor is likely to invade important blood vessels during the subsequent study;
9. Those allergic to the use of drugs or their ingredients in this regimen;
10. Grade 2 peripheral neurological disease or hearing loss according to the criteria of common adverse event terms (NCI CTCAE V5.0);
11. Pregnant or lactating women;
12. Patients with a history of psychiatric substance abuse and unable to quit or with mental disorders;
13. The investigator is not considered fit to join the investigator; Unwilling to participate in the study or unable to sign the informed consent form

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFSProgression-Free-Survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin MM GE, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No